CLINICAL TRIAL: NCT07043296
Title: Risk Factors for Deep Sternal Wound Infection After Coronary Artery Bypass Grafting
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Alaa Eldien Ali Hassan, residant doctor at Assiut university, Assiut University
Other Study IDs: DSWI risk factors
Record Dates: First submitted 2025-06-20; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Coronary Artery Bypass Grafting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: patients for CABG operation

SUMMARY:
Deep sternal wound infection (DSWI) constitutes a serious complication after coronary artery bypass grafting (CABG) surgery with potentially devastating consequences for patients. (1) Although median sternotomy is known to offer an excellent approach in CBAG, the impact of DSWI on patient prognosis remains significant. (2) The advances made in the field of prevention allowed the incidence of DSWI to decrease drastically in CBAG operations. (3,4) DSWI has been shown to lead to life- threatening complications linked with an increase in long and short-term mortality, morbidity, cost of care, prolonged hospital stays and in-hospital mortality. (5-8) There are a reported numerous risk factors potentially contributing to the development of DSWI in CABG, including the use of the internal thoracic artery for revascularization, long operative time, reoperation, an excessive use of bone wax and electrocoagulation, peripheral mechanical ventilation and other patient- related immunosuppressive risk factors. (9,10) Metabolic disorders such as diabetes, hypertension, dyslipidaemia and obesity leading to increased risk of poor clinical outcomes. (11) The aim of this study is determine the cut off point for some of known risk factors for deep sternal wound infection after Coronary artery bypass grafting.

ELIGIBILITY:
Inclusion Criteria:

* All patients for CABG operation

Exclusion Criteria:

* patients who died during operations or shortly after it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients for CABG operation
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
postoperative infection | 30 DAy
  postoperative wound infection after CABG